CLINICAL TRIAL: NCT00743327
Title: Metabolic and Cardiovascular Complications in Men With Prostate Cancer Undergoing Long-term Androgen Deprivation Therapy
Brief Title: Androgen Deprivation Therapy Study
Acronym: ADT
Status: Terminated | Type: Observational
Why Stopped: No Participants completed study
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: AG0107
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Hypogonadism; Metabolic Syndrome; Diabetes; Inflammation
Keywords: hormone therapy
MeSH Terms: conditions — Hypogonadism; Metabolic Syndrome; Diabetes Mellitus; Inflammation | interventions — Pioglitazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Muscle biopsy specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Participants receiving ADT and pioglitazone
  Interventions: Drug: Pioglitazone
- 2: Participants receiving ADT only
- 3: Participants not receiving ADT and in remission from prostate cancer

INTERVENTIONS:
Drug: Pioglitazone — 45mg capsule, once daily for 1 year
  Other Names: Actos
  Groups: 1

SUMMARY:
The purpose of this study is to examine the link between low testosterone and insulin resistance/diabetes in men undergoing androgen deprivation therapy for prostate cancer. The study will also evaluate other cardiovascular risk factors in these men.

DETAILED DESCRIPTION:
Lowering of testosterone levels, by medications or surgery (Androgen Deprivation Therapy or ADT), is commonly used in the treatment of prostate cancer. The adverse effects of low testosterone include decreased sex drive, impotence, decreased lean body mass and muscle strength, increased fat mass, decreased quality of life and osteoporosis.

An increase in body fat and decrease in lean body mass may contribute to a decrease in the body's ability to use insulin effectively, leading to insulin resistance and diabetes. Low testosterone levels are also associated with elevated total cholesterol, LDL-cholesterol and triglycerides.

Two groups of non-diabetic men will be studied:

1. Men with known history of prostate cancer who were treated with surgery and/or radiation therapy and are now in remission and not receiving androgen deprivation therapy (non-ADT group).
2. Men with newly diagnosed or known history of prostate cancer who are being advised by their physicians to begin androgen deprivation therapy (ADT group).

The non-ADT group and half of the ADT group will be observed for the development of insulin resistance/diabetes. The other half of the ADT group will receive a diabetes medication called Pioglitazone (Actos) to evaluate any beneficial effects of this medication in the prevention of metabolic dysfunction.

The study will consist of a screening visit and 6 additional study visits throughout one year. Procedures during this study include blood draws, MRI, CT, DEXA scan, insulin clamp procedures, oral glucose tolerance tests, carotid IMT, pulse wave velocity, neuropsychological testing, physical exams and an optional muscle biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Men 18 years of age or older with prostate cancer
* Planning to undergo long-term (at least 12 months) ADT
* No known history of diabetes
* No history of ADT

Exclusion Criteria:

* History of ADT or any prior diagnosis of hypogonadism
* Fasting glucose or oral glucose tolerance test results in the diabetic range
* Heart failure (NY classification III or IV)
* Testosterone level less than 250 ng/dl on screening
* History of heart attack or open-heart surgery within the past 6 months
* Use of steroids within the past 3 months, including prednisone, cortisone injections, inhaled steroids (topical steroids are acceptable)
* Use of anabolic steroids (testosterone, DHEA, DHEAS) or any growth promoters (growth hormone itself or analogs of growth hormone) in the past 12 months
* Liver function tests more than 3 times upper normal limits
* Undergoing intermittent ADT
* Uncontrolled thyroid disease (hyper- or hypo-thyroidism)
* Anemia, defined as hematocrit less than 38%
* Not physically capable of completing the tests

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample of men ages 18 and older with prostate cancer
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Evaluation for the development of incident diabetes | every 3 months

SECONDARY OUTCOMES:
Evaluation for other cardiovascular risk factors, markers of inflammation and immunological changes | every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Josephine M. Egan, MD, Principal Investigator — National Institute on Aging, Intramural Research Program
Locations (1):
- NIA Clinical Research Unit located at Harbor Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Dockery F, Bulpitt CJ, Agarwal S, Donaldson M, Rajkumar C. Testosterone suppression in men with prostate cancer leads to an increase in arterial stiffness and hyperinsulinaemia. Clin Sci (Lond). 2003 Feb;104(2):195-201. doi: 10.1042/CS20020209. PMID 12546642
- [Background] Smith MR, Lee H, Nathan DM. Insulin sensitivity during combined androgen blockade for prostate cancer. J Clin Endocrinol Metab. 2006 Apr;91(4):1305-8. doi: 10.1210/jc.2005-2507. Epub 2006 Jan 24. PMID 16434464
- [Background] Basaria S, Muller DC, Carducci MA, Egan J, Dobs AS. Hyperglycemia and insulin resistance in men with prostate carcinoma who receive androgen-deprivation therapy. Cancer. 2006 Feb 1;106(3):581-8. doi: 10.1002/cncr.21642. PMID 16388523
- [Background] Keating NL, O'Malley AJ, Smith MR. Diabetes and cardiovascular disease during androgen deprivation therapy for prostate cancer. J Clin Oncol. 2006 Sep 20;24(27):4448-56. doi: 10.1200/JCO.2006.06.2497. PMID 16983113
- [Background] Braga-Basaria M, Dobs AS, Muller DC, Carducci MA, John M, Egan J, Basaria S. Metabolic syndrome in men with prostate cancer undergoing long-term androgen-deprivation therapy. J Clin Oncol. 2006 Aug 20;24(24):3979-83. doi: 10.1200/JCO.2006.05.9741. PMID 16921050